CLINICAL TRIAL: NCT01962779
Title: Sleep, Aging and Risk for Alzheimer's Disease (SARA) Study
Brief Title: Sleep, Aging and Risk for Alzheimer's Disease
Acronym: SARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-03068; R01HL118624 (NIH)
Record Dates: First submitted 2013-08-27; First posted 2013-10-14 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Sleep Disordered Breathing; Alzheimer's Disease
Keywords: Sleep Disordered Breathing; Cognitively normal elderly; Alzheimer's disease; Prevention; Continuous positive airway pressure (CPAP)
MeSH Terms: conditions — Sleep Apnea Syndromes; Alzheimer Disease | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous positive airway pressure (Experimental): Moderate to severe SDB subjects will be offered a 6-month therapy with continuous positive airway pressure (CPAP).
  Interventions: Other: Continuous positive airway pressure (CPAP)
- No intervention (No Intervention): Subjects that refuse treatment with CPAP or that have a poor long-term compliance will be considered controls.

INTERVENTIONS:
Other: Continuous positive airway pressure (CPAP) — Continuous positive airway pressure (CPAP). CPAP typically is used for people who have breathing problems, such as sleep apnea.
  Arms: Continuous positive airway pressure

SUMMARY:
Our preliminary data show for in cognitively-normal elderly, that Sleep Disordered Breathing (SDB) is associated with the increase of cerebrospinal fluid (CSF) phosphorylated-Tau (P-Tau) and total-Tau (T-Tau), decreases in medial temporal lobe glucose uptake (FDG-PET) and volume (MRI) and progressive memory decline, all of which have been shown to be useful in predicting future dementia in older adults. These findings raise the question as to whether Alzheimer's disease (AD) tissue damage causes SDB in the elderly, or alternatively, if SDB acts as a risk factor for AD neurodegeneration. In the proposed study, we will investigate these mechanistic hypotheses in cognitively normal elderly by examining the longitudinal associations between SDB and cognitive decline, novel MR neuroimaging and CSF biomarkers for neurodegeneration; while our secondary goal is to launch a pilot treatment study to aid in interpreting the mechanistic hypotheses and to examine the effects of nasal continuous positive airway pressure (CPAP) on cognitive decline and neurodegeneration.

DETAILED DESCRIPTION:
Sleep disordered breathing (SDB) is a common disorder with an estimated prevalence in the elderly ranging from 30-80%. The relevance of this high frequency in late life is emerging, as recent evidence suggests that SDB may be associated with the development of mild cognitive impairment and dementia. Alzheimer's disease (AD) is the most common form of dementia and affects nearly 45% of the population older than 85. Hippocampal atrophy and glucose hypometabolism, as well as changes in cerebrospinal fluid (CSF) levels of amyloid beta-42 (Aβ42), phosphorylated-tau (P-Tau) and total-tau (T-Tau), have been shown to be useful in predicting future decline in cognitively normal older adults, which suggests that AD pathology is detectable prior to cognitive impairment in at-risk subjects. This "presymptomatic phase", in which tissue damage is minimal and whose detection precedes clinical symptoms, is an ideal stage for risk factor analysis and intervention trials. Our preliminary data show, for the first time in cognitively-normal elderly, that the severity of SDB (as measured by respiratory events with 4% desaturation, Apnea Hypopnea Index 4% [AHI4%]) is associated with the increase of CSF P-Tau and T-Tau, a decrease in glucose uptake (measured by FDG-PET) in the medial temporal lobe, reduced hippocampal volume, and longitudinal memory decline. These findings raise the question as to whether AD tissue damage causes SDB in the elderly, or alternatively, if SDB acts as a risk factor for neurodegeneration. The proposed parent grant for this project conducted at the NYU Center for Brain Health (CBH), is a 5-year NIH-funded longitudinal study of 180 normal elderly (50-95 years), who will undergo complete baseline and 24 month follow-up evaluations. The exams include MR imaging: both structural and cerebral blood flow (CBF) using a novel NYU arterial spin labeling (ASL) protocol and regional brain vasoreactivity estimates after CO2 breathing (VR-CO2); as well as both plasma and CSF biomarkers. The present ancillary proposal, performed in collaboration with NYU's Sleep Disorders Center, will investigate: 1) SDB as a longitudinal predictor of changes in memory, levels of P-tau and T-Tau, hippocampal atrophy, and the blunted VR-CO2 response (all these effects of SDB were observed in cross-section in our pilot work); and 2) if these SDB related phenomena in normal elderly are susceptible to intervention with nasal continuous positive airway pressure (CPAP) in moderate-to-severe SDB subjects. This study has the potential to identify: 1) a highly prevalent AD-related mechanism by which SDB contributes to cognitive decline; 2) the alternative hypothesis, the presence of biomarker features of AD as risks factors for SDB; and 3) that the treatment of SDB with CPAP improves cognition through an AD-related pathway in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with normal cognition and >50 years of age will be enrolled. Younger subjects are not included as the risk for cognitive impairment is too low. Moreover, by selecting this age-range we minimize the possibility of including early-onset genetic forms of neurodegenerative diseases such as Alzheimer's disease and Frontotemporal Dementia.
* Normal subjects will be within normal limits on neurological and psychiatric examinations. All subjects enrolled will have both a Clinical Dementia Rating = 0 and Global Deterioration Scale < 3.
* All subjects will have had a minimum of 12 years education.The education restriction reduces performance variance on cognitive test measures and improves the sensitivity for detecting pathology and disease progression using the robust norms available at NYU School of Medicine.
* All subjects will have an informed family member or life partner interviewed to confirm the reliability of the subject interview. All subjects will agree to the MRI imaging, the lumbar puncture, apolipoprotein E (ApoE) genotyping and DNA banking

Exclusion Criteria:

* Diagnosis of any brain disease or MRI evidence of brain damage including significant trauma, hydrocephalus, seizures, mental retardation or other serious neurological disorder (e.g. Parkinson's disease or other movement disorders). Persons with silent cortical infarcts are excluded. Subcortical infarcts and white matter lesions are not exclusions.
* History of brain tumor.
* Any radiation or chemotherapy anywhere in the body in the past 3-years.
* Significant history of alcoholism or drug abuse.
* History of psychiatric illness (e.g., schizophrenia, mania, PTSD, or life long history of major depression).
* Hamilton Depression Scale >16 only with history of life long depressive episodes. Otherwise not excluded.
* Evidence of clinically relevant and uncontrolled cardiac, pulmonary, or hypothyroid or hematological conditions. Insulin dependent diabetes and/or history or treated hypertension are not an exclusion. Normal subjects with current levels of HbA1c >5.9% or diabetics >7.0% (American Diabetes Association, 2010) and/or current blood pressure levels >140/90 mm Hg (JNC on Prevention, Detection, Evaluation and Treatment of High Blood Pressure, 2003) will be advised to seek referral.
* Physical impairment of such severity as to adversely affect the validity of psychological testing.
* Hostility or refusal to cooperate.
* Any prosthetic devices (e.g., pacemaker or surgical clips) that constitutes a hazard for MRI imaging.
* History of a first-degree family member with early onset (before age 65) dementia.
* Medications adversely affecting cognition will result in exclusion. The excluded medications include:

  * Antidepressants with anti-cholinergic properties.
  * Regular use of narcotic analgesics (>2 doses per week).
  * Use of neuroleptics with anti-cholinergic properties.
  * Other medications with central nervous system anticholinergic activity.
  * Use of Anti-Parkinsonian medications.
* At the baseline individuals taking physician ordered or off-label memory or other cognitive enhancing medications (e.g. cholinesterase inhibitors or memantine) are excluded. At the follow-up these medications are allowed. Also excluded at baseline are individuals taking physician ordered, but off-label memory enhancements. Individuals taking over the counter memory enhancing or protecting medications (e.g. ginkgo biloba, vitamins) are not excluded.
* Patients with significant physical changes (e.g. amputations or loss of sensory input) as these may affect the MRI blood flow measures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Observational. Cerebrospinal fluid (CSF) biomarkers of risk for Alzheimer's disease (AD) in sleep disordered breathing (SDB) subjects. | Baseline
  At cross section, levels of CSF P-Tau, T-Tau and Aβ42 (in pg/mL) in subjects with SDB
Observational. Structural MRI hippocampal volume in SDB subjects. | Baseline
  At cross section, hippocampal volume (in mm3) in subjects with SDB
Observational. MRI-ASL vasoreactivity response to CO2 challenge in subjects with SDB | Baseline
  At cross-section, MRI-ASL measured vasoreactivity responses to CO2 (% of brain vasoreactivity to hypercapnia) in subjects with SDB

SECONDARY OUTCOMES:
Interventional CPAP Clinical Trial, memory changes after CPAP treatment | Change from baseline in memory tests at 6 months
  All subjects with moderate-to-severe SDB (Apnea Hypopnea Index with 4% desaturation >15) will be prescribed 6-month treatment with CPAP. Changes after treatment in declarative memory (measured using tests from the Wechsler and Guild Memory scales from our neuropsychological battery) at 6 months.
Interventional CPAP Clinical Trial, CSF biomarker changes after CPAP treatment | Change from baseline in CSF biomarkers at 6 months
  All subjects with moderate-to-severe SDB (Apnea Hypopnea Index with 4% desaturation >15) will be prescribed 6-month treatment with CPAP. Change after a 6 month treatment in CSF levels of P-Tau (pg/mL), T-Tau (pg/mL) and Aβ42 (pg/mL)
Interventional CPAP Clinical Trial, MRI biomarker changes | Change from baseline in MRI biomarkers at 6 months
  All subjects with moderate-to-severe SDB (Apnea Hypopnea Index with 4% desaturation >15) will be prescribed 6-month treatment with CPAP. Changes after a 6 month treatment in brain vasoreactivity response to CO2 (measured by % of vasoreactivity response to hypercapnia) and hippocampal volume in mm3

OTHER OUTCOMES:
Observational. 2-year longitudinal cognitive memory outcomes | Change from baseline in memory tests at 24 months
  Changes in memory (tests from the Wechsler and Guild Memory scales from our cognitive battery) in SDB-at-baseline subjects (non-treated with CPAP) at the 2-year follow-up
Observational. 2-year longitudinal AD-biomarker CSF outcomes | Change from baseline in CSF biomarkers at 24 months
  Changes in CSF P-Tau levels, T-Tau (pg/mL) and Aβ42(pg/mL) in SDB-at-baseline subjects (non-treated with CPAP) at the 2-year follow-up
Observational. 2-year longitudinal MRI structural and functional outcomes | Change from baseline in MRI biomarkers at 24 months
  Changes in hippocampal atrophy (mm3) and VR-CO2 responses (% of vasoreactivity response to hypercapnia) in SDB-at-baseline subjects (non-treated with CPAP) at the 2-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo S Osorio, MD, Principal Investigator — Research Assistant Professor
Locations (2):
- United States (2):
  - NYU Sleep Disorders Center, New York, New York
  - NYU Center for Brain Health, New York, New York

REFERENCES:
- [Derived] Osorio RS, Ducca EL, Wohlleber ME, Tanzi EB, Gumb T, Twumasi A, Tweardy S, Lewis C, Fischer E, Koushyk V, Cuartero-Toledo M, Sheikh MO, Pirraglia E, Zetterberg H, Blennow K, Lu SE, Mosconi L, Glodzik L, Schuetz S, Varga AW, Ayappa I, Rapoport DM, de Leon MJ. Orexin-A is Associated with Increases in Cerebrospinal Fluid Phosphorylated-Tau in Cognitively Normal Elderly Subjects. Sleep. 2016 Jun 1;39(6):1253-60. doi: 10.5665/sleep.5846. PMID 26951396